CLINICAL TRIAL: NCT04971031
Title: A Multi-Center Randomized, Double-Masked, Parallel Design, Vehicle-Controlled Phase 2 Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: A Clinical Trial to Assess Subjects With Dry Eye Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-024
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) administered 7 times over two consecutive days. (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle Ophthalmic Solution administered 7 times over two consecutive days. (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered 7 times over two consecutive days.
  Arms: Reproxalap Ophthalmic Solution (0.25%) administered 7 times over two consecutive days.
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution administered 7 times over two consecutive days.
  Arms: Vehicle Ophthalmic Solution administered 7 times over two consecutive days.

SUMMARY:
A Multi-Center Randomized, Double-Masked, Parallel Design, Vehicle-Controlled Phase 2 Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects with Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age (either gender and any race);
2. Reported history of dry eye for at least 6 months prior to Visit 1;
3. Reported history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1.

Exclusion Criteria:

1. Clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
2. Diagnosis of an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
3. Contact lens use within 7 days of Visit 1 or anticipate using contact lenses during the trial;
4. Eye drop use within 2 hours of Visit 1;
5. Previous laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
6. Cyclosporine 0.05% or 0.09% or lifitegrast 5.0% ophthalmic solution use within 90 days of Visit 1;
7. Be receiving systemic corticosteroid therapy (not including inhaled corticosteroids) within 14 days of Visit 1 or anticipate such therapy throughout the study period;
8. Planned ocular and/or lid surgeries over the study period or any ocular surgery within 6 months of Visit 1;
9. Temporary punctal plugs during the study that have not been stable within 30 days of Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred fifty-eight subjects were randomized in the trial.
Groups:
- Reproxalap (0.25%): Reproxalap ophthalmic solution administered 7 times over two consecutive days
- Vehicle: Vehicle ophthalmic solution administered 7 times over two consecutive days
Period: Overall Study
Arm/Group | Reproxalap (0.25%) | Vehicle
Started | 80 | 78
Completed | 79 | 75
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproxalap (0.25%) | Vehicle | Total
Number analyzed (Participants) | 80 | 78 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 48 | 91
  >=65 years | 37 | 30 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 55 | 114
  Male | 21 | 23 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 11 | 16
  Not Hispanic or Latino | 75 | 67 | 142
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 3 | 5
  Black or African American | 8 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 67 | 68 | 135
  Other | 0 | 1 | 1
  Multiple | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 80 | 78 | 158
Iris Color (Right Eye) [Count of Participants; unit: Participants]
  Black | 0 | 0 | 0
  Blue | 18 | 18 | 36
  Brown | 44 | 31 | 75
  Hazel | 7 | 17 | 24
  Green | 11 | 12 | 23
  Gray | 0 | 0 | 0
  Other | 0 | 0 | 0
Iris Color (Left Eye) [Count of Participants; unit: Participants]
  Black | 0 | 0 | 0
  Blue | 18 | 18 | 36
  Brown | 44 | 31 | 75
  Hazel | 7 | 17 | 24
  Green | 11 | 12 | 23
  Gray | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Redness Assessed Via Digital Photography Over 90 Minutes in the Dry Eye Chamber
Description: Change from baseline comparison of reproxalap to vehicle for conjunctival redness on a 0 to 4 scale ( 0 = normal, 4 = prominent), where a high score means a worse outcome. The intervention was administered bilaterally. The least squares mean (standard error) was derived from mixed model repeated measure for change from baseline included baseline, treatment group, and nominal time point as fixed effects.
Time Frame: The efficacy assessment period was assessed during the 90-minute dry eye chamber at Day 2; baseline was Pre-Dose #1 at Day 1.
Population: Intent-to-Treat Population with observed data only
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reproxalap (0.25%) | Vehicle
Number analyzed (Participants) | 80 | 78
units on a scale | 0.066 (0.0346) | 0.183 (0.0353)

2. Primary Outcome: Subject-reported Ocular Dryness Score (0 - 100 Visual Analogue Scale (VAS))
Description: Change from baseline comparison of reproxalap to vehicle for subject-reported ocular dryness score VAS (0 = no discomfort, 100 = maximal discomfort), where a high score means a worse outcome. The intervention was administered bilaterally. The least squares mean (standard error) was derived from mixed model repeated measure for change from baseline included baseline, treatment group, and nominal time point as fixed effects.
Time Frame: as for outcome 1
Population: Intent-to-Treat Population with observed data only
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reproxalap (0.25%) | Vehicle
Number analyzed (Participants) | 80 | 78
units on a scale | -5.7 (2.44) | -3.8 (2.51)

3. Primary Outcome: Schirmer Test Change From Baseline After the First Dose on Day 1
Description: Change from baseline comparison of reproxalap to vehicle for Schirmer test on a millimeter line (0 = none, 35 = maximum), where a shorter length indicates a worse outcome. The intervention was administered bilaterally. The least squares mean (standard error) was derived from mixed model repeated measure for change from baseline included baseline and treatment group as fixed effects.
Time Frame: The efficacy assessment period was before and after the final dose on Day 1; baseline was Pre-Dose #1 at Day 1.
Population: Intent-to-Treat Population with observed data only
Measure: Least Squares Mean (Standard Error); unit: length in millimeters
Arm/Group | Reproxalap (0.25%) | Vehicle
Number analyzed (Participants) | 80 | 78
length in millimeters | 4.2 (0.83) | 2.1 (0.84)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately one week.
Description: There were 158 subjects randomized in the trial (Intent-to-treat population). There were 156 subjects exposed to study drug (Safety population). Collection of adverse events is based on the Safety population.
Arm/Group | Reproxalap (0.25%) | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/77
Other Adverse Events (participants affected / at risk) | 52/79 | 3/77
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap (0.25%) (N=79) | Vehicle (N=77)
General disorders and administration site conditions (General disorders) | 52 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT04971031/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT04971031/SAP_001.pdf